CLINICAL TRIAL: NCT02523508
Title: Does Passive Spinal Mobilization Improve Lower Limbs Strength and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LO CHI NGAI, Clinical Associate, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20150310003
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Passive manual lumbar mobilization on L2-3 level
  Interventions: Behavioral: Experimental group
- Control group (Placebo Comparator): Passive limb mobilization which did not involve the spine
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Experimental group — Subject will be put into lying position, small amplitude of passive movement on the lumbar spine of the subject. The procedure will last for 1 minute.
  Arms: Experimental group
Other: Control group — Passive limb mobilization which did not involve the spine
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Previous studies have shown that peripheral muscles weakness or inhibition is related to spinal disorders. Passive mobilization and manipulation are likely to reverse such muscle weakness. The purpose of the study was to assess the effect of spinal mobilization on the maximal muscle strength of the hip flexors and motor function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults have no active back or hip pain

Exclusion Criteria:

* Subjects with active back or hip pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hip flexor strength | 10 minutes after the intervention
  The hip flexor strength measured by the hand-held dynamometer

SECONDARY OUTCOMES:
Running speed | 10 minutes after the intervention
  The running time for a 100-meter distance

CONTACTS AND LOCATIONS:
Overall Officials: Chi Ngai Lo, Master, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No